CLINICAL TRIAL: NCT02407379
Title: Photoablative-photodynamic (PAPD) Diode Laser Therapy Adjunctive to Scaling and Root Planing in Periodontitis
Brief Title: Diode Laser and SRP in Chronic Periodontitis
Acronym: PAPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odontostomatologic Laser Therapy Center, Florence, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: OLTC014
Record Dates: First submitted 2014-07-09; First posted 2015-04-03 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Periodontitis
Keywords: Laser; periodontitis; scaling root planing; bacteria; PMN
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAPD+SRP Quadrant (Active Comparator): This quadrant, randomly selected in each patients, undergoes treatment with PAPD+ SRP
  Interventions: Procedure: PAPD+SRP
- Sham-laser + SRP (Sham Comparator): This quadrant, randomly selected in each patients, undergoes treatment with sham-laser + SRP
  Interventions: Procedure: Sham-laser +SRP

INTERVENTIONS:
Procedure: PAPD+SRP — Photoablation of the gingival epithelium was performed with at 810 nm diode laser (1 W output power, continuous wave mode, 66.7 J/cm2, a 0.6 mm optical fiber). SRP was performed using curettes. The periodontal tissues and the dental root were rinsed with the photosensitizer agent methylene blue (0.3% w/v in water). After 5 min., the treated areas were irradiated with at 635 nm diode laser (100 mW output power, continuous wave mode, 0.6 mm optic fiber). The photodynamic treatment was repeated once weekly until normalization of the cytodiagnostic parameters (range: 4-10 applications).
  Arms: PAPD+SRP Quadrant
Procedure: Sham-laser +SRP — Sham-treatment was similar to the previously described treatment but with switched off laser, followed by scaling and root planing
  Arms: Sham-laser + SRP

SUMMARY:
The purpose of this study is to compare the efficacy of photoablative and photodynamic diode laser in adjunct to scaling-root planing (PAPD+SRP) and SRP alone for the treatment of periodontitis.

DETAILED DESCRIPTION:
The present study is a randomized, blinded, controlled clinical trial, which used a split-mouth design. All patients were informed individually about the nature of the proposed treatment, and informed consent forms were signed. Twenty-four patients were studied. Maxillary left or right quadrants were randomly assigned to PAPD laser treatment or sham-treatment and SRP. PAPD consisted of: i) photoablative gingival epithelium with diode laser (λ 810 nm, 1 W); ii) photodynamic treatments (4-10 weekly) with diode laser (λ 635 nm, 100 mW) and 0.3% methylene blue as photoactive antiseptic, performed after SRP. Sham-treatment was similar but with switched off laser.

Efficacy evaluations, including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP) was performed at baseline ,1year, and year 3 using a conventional manual periodontal probe. Polymorphonuclear leukocytes (PMN), erythrocytes (RBC), damaged epithelial cells (DEC) and bacteria were assayed by cytofluorescence on gingival exfoliative samples at baseline, 6 month and 1, 3, 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Periodontitis:Presence of at least two teeth with at least one site with pocket probing depth (PD) ranging from 4 to 10 mm in each upper maxillary quadrant and with bleeding on probing (BOP)
2. A minimum of five natural teeth in each studied quadrant.

Exclusion Criteria:

1. History of systemic diseases (diabetes mellitus, cancer, HIV, metabolic and endocrine diseases)
2. Pregnancy or lactation
3. Chronic high-dose steroid use
4. Previous or current radiation or immunosuppressive therapies
5. Ongoing orthodontic treatments
6. Extensive carious lesions
7. Recurrent antibiotic medications during the 6 months preceding the study
8. Class III tooth mobility
9. Heavy contamination by spirochetes and fungal pathogens on tongue and oral mucosa

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
PD | baseline, 1 year
  Change in probing pocket depth

SECONDARY OUTCOMES:
CAL | baseline, 1 year
  Change in mean attachment level
BoP | baseline, 1 year
  Change in mean bleeding on probing
PMN, DEC, bacteria | baseline, 1 year
  Change in mean additional disease markers, namely polymorphonuclear leukocytes (PMN), erythrocytes (RBC), damaged epithelial cells (DEC) and bacteria were assayed by cytofluorescence on gingival exfoliative samples.
Patient-reported outcomes | baseline, 1 year
  Individual evaluation of pain/discomfort assessed by a visual analogue score interview

CONTACTS AND LOCATIONS:
Overall Officials: Marco Giannelli, Principal Investigator — Odontostomatologic laser therapy center
Locations (1):
- Odontostomatologic laser therapy center, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giannelli M, Materassi F, Fossi T, Lorenzini L, Bani D. Treatment of severe periodontitis with a laser and light-emitting diode (LED) procedure adjunctive to scaling and root planing: a double-blind, randomized, single-center, split-mouth clinical trial investigating its efficacy and patient-reported outcomes at 1 year. Lasers Med Sci. 2018 Jul;33(5):991-1002. doi: 10.1007/s10103-018-2441-9. Epub 2018 Jan 18. PMID 29349511